CLINICAL TRIAL: NCT06155006
Title: Adult Screening for Hepatitis c and Linkage to Treatment in Hospitals in Colombia
Acronym: HCVLINKAGE
Status: Recruiting | Type: Observational
Sponsor: Asociación Colombiana de Hepatología (Other)
Collaborators: Hospital Pablo Tobón Uribe (Other)
Responsible Party: Principal Investigator, Diana Rocio Chavez Bejarano, Epidemiology, Asociación Colombiana de Hepatología
Other Study IDs: CO-US-987-6934; CO-US-987-6934 (Other Grant/Funding Number: Colombian Association of Hepatology)
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Hepatitis C Virus Infection
Keywords: prevalence; rapid diagnostic tests
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with risk factors for hepatitis C virus: All persons over 18 years of age who are treated in the included health care institutions (IPS) and who are users of hospitalization, emergency, outpatient, and any other hospital care services.
  Interventions: Diagnostic Test: rapid diagnostic test HCV Ab Plus Rapid test

INTERVENTIONS:
Diagnostic Test: rapid diagnostic test HCV Ab Plus Rapid test — The sample will be taken by trained personnel by capillary puncture of the thumb region of the fingers of the right hand, after asepsis and antisepsis, the rapid diagnostic test HCV Ab Plus Rapid test with INVIMA registration 2018RD-0002353-R1 will be used with operational characteristics that allow its performance at the point of care obtaining a result in 15 to 20 minutes. This rapid test for antibodies against HCV may be replaced by another test with similar operational characteristics (sensitivity and specificity).
  Other Names: Opportunity screening

SUMMARY:
Introduction: Hepatitis C virus infection is a major cause of chronic hepatitis, cirrhosis, and liver cancer. The risk of developing cirrhosis for people with chronic infection with the virus ranges from 15% to 30% over a 20-year period. According to 2019 data from the World Health Organization there are 58 million people living with chronic hepatitis C infection. Three-quarters of those infected live in low- to middle-income countries, some of which lack budgets for screening, diagnosis and treatment campaigns. While good progress has been made in several countries, a significant gap in testing and treatment remains. Barriers to timely diagnosis include lack of awareness on the part of health professionals, availability and access to screening tests. Simplifying the cascade of care for this pathology would help ensure that more patients remain involved in the care pathway and ultimately achieve global goals.

Objective: To estimate the prevalence of anti-HCV antibodies in patients with risk factors for hepatitis C virus captured by opportunity screening in the included hospital institutions.

Methodology: Descriptive multicenter cross-sectional study. A total of 27160 participants among the seven institutions, 3880 per institution. Includes all persons over 18 years of age attended in the included health service provider institutions (IPS) who are users of hospitalization, emergency, outpatient and any other hospital care services. Application of a questionnaire to identify the inclusion criteria and data collection, signature of informed consent, sample collection by rapid test Abbott HCV rapid test - BIOLINE HCV and evaluation by tele-consultation by hepatologist principal investigator who will guide you to access the confirmatory test for HCV (viral load for Hepatitis C), the study will assume responsibility for its realization.

DETAILED DESCRIPTION:
Research question

¿What is the prevalence of HCV in the population with risk factors for hepatitis C virus infection captured by screening with rapid tests in health care institutions in Colombia?

Through this observational, multicenter, hospital population study, the prevalence will be determined by screening patients with risk factors for hepatitis C by rapid antibody test, to subsequently perform confirmation with viral load PCR in those seropositive. In addition, support will be provided to patients to facilitate their treatment adherence.

The benefits would be related to raising awareness of the importance of the active search for these patients, reducing the health impact for the screened population, incorporating these strategies in the country's hospital institutions, and obtaining epidemiological information that helps to understand the magnitude of the disease and the opportunity for its elimination.

ELIGIBILITY:
Inclusion Criteria:

Have at least one of the following risk factors for hepatitis C.

* Over 50 years of age with no risk factors.
* Over 18 years old and less than 50 years old with risk factors for hepatitis C. Persons who have received medical or dental interventions in health care settings.

Persons who have had tattoos, body piercings, or scarification procedures. Persons with HIV or hepatitis B infection. Persons who inject drugs. Persons who have used intranasal drugs. Persons deprived of liberty and previously incarcerated persons. Anyone with abnormal liver tests or liver disease. Students, health care workers, or members of public safety (e.g. correctional service officers or police) who have come into contact with blood at work through needlestick or sharps injuries. Anyone who has undergone hemodialysis. Persons who received transfusions in Colombia before 1996. Persons with comorbidities potentially associated with CH: diabetes, ischemic heart disease, cryoglobulinemia, chronic renal failure, Sjögren's syndrome, hypothyroidism, lichen planus, rheumatoid arthritis, HIV, non-Hodgkin's lymphoma, acute lymphoblastic leukemia, waldenstrom's macroglobulinemia.

* Individuals previously treated for HCV with sustained viral response in whom reinfection is suspected (individuals who continue to engage in risk behaviors)
* Accept to participate in the study by signing the informed consent form.

Exclusion Criteria:

* Have or have had hepatitis C with a proven cure by viral load at 12 weeks after the end of treatment without risk behaviors for reinfection.
* Be on antiviral treatment against chronic hepatitis C virus.
* That the patient voluntarily and consciously refuses to sign the informed consent form or is unable to give it due to any type of physical and/or mental disability.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All persons over 18 years of age who are treated in the included health care institutions (IPS) and who are users of hospitalization, emergency, outpatient, and any other hospital care services.
Sampling Method: Non-Probability Sample
Enrollment: 25669 (Estimated)
Dates: Start 2023-12-16 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence | 12 months
  Hepatitis C virus prevalence

SECONDARY OUTCOMES:
Opportunity for treatment | 12 months
  Access to treatment for hepatitis C virus infection

CONTACTS AND LOCATIONS:
Overall Officials: Javier Hernández Blanco, MD, Study Director — Asociación Colombiana de Hepatología
Locations (2):
- Colombia (2):
  - Hospital Pablo Tobón Uribe, Medellín, Antioquia
  - Hospital Universitario Julio Méndez Barreneche E.S.E., Santa Marta, Magdalena Department

IPD SHARING:
Plan to Share IPD: No
Informed consent will be requested in written form to all participants, giving clear and easily understandable information about the objectives of the research. The consent will be explained and doubts about it will be resolved and complete freedom of withdrawal of consent will be given at any time during the study, for the reasons that the subject considers.
  The study will be coordinated by health professionals and the sampling and data collection will be performed by nursing assistants trained in rapid tests. The confidentiality of the data collected will be guaranteed, the information obtained will not be used for purposes other than the current research process, and sensitive data or data that allow the identification of the participating individuals will not be published when the information is disclosed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT06155006/Prot_SAP_000.pdf